CLINICAL TRIAL: NCT01111890
Title: Comparison of the Efficacy of AZARGA® Versus COSOPT® in Patients With Open-Angled Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-09-17
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2012-01

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Azarga; brinzolamide; dorzolamide-timolol combination; dorzolamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azarga (Experimental): Azarga (brinzolamide 1% / timolol 0.5%)
  Interventions: Drug: Azarga (brinzolamide 1% / timolol 0.5%)
- Cosopt (Active Comparator): Cosopt (dorzolamide 2% / timolol 0.5%)
  Interventions: Drug: Cosopt (dorzolamide 2% / timolol 0.5%)

INTERVENTIONS:
Drug: Azarga (brinzolamide 1% / timolol 0.5%) — Dosed twice daily at 9:00 AM and 9:00 PM for 12 weeks
  Arms: Azarga
Drug: Cosopt (dorzolamide 2% / timolol 0.5%) — Dosed twice daily at 9:00 AM and 9:00 PM for 12 weeks
  Arms: Cosopt

SUMMARY:
Subjects are dosed twice daily at 9AM and 9PM for 12 weeks. The primary efficacy variable is the mean change in Intraocular Pressure (IOP) from baseline to 12 weeks. Secondary efficacy variable: % IOP ≤ 18 millimeters mercury (mmHg). Exploratory endpoint: Ocular discomfort scale after first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years of age.
2. Must have a clinical diagnosis of ocular hypertension, primary open-angle or pigment dispersion glaucoma in at least one eye (study eye).
3. Must have IOP considered to be safe, in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
4. Must be willing to discontinue the use of all other ocular hypotensive agents prior to receiving the assigned study drug at Visit 1, throughout the study period.
5. Must have an IOP of between 19 to 35 mmHg in at least one eye (which would be the study eye).
6. For the eyes not included in the study, the intraocular pressure should be able to be controlled on no pharmacologic therapy or on the study medicine alone.

Exclusion Criteria:

1. Known medical history of allergy, hypersensitivity or poor tolerance to any components of the preparations to be used in this study that is deemed clinically significant in the opinion of the Principal Investigator.
2. Presence of other primary or secondary glaucoma not listed in inclusion criterion #2.
3. Any abnormality preventing reliable applanation tonometry in study eye(s).
4. Risk of visual field or visual acuity worsening due to participation in the study, in the investigator's best judgment.
5. Progressive retinal or optic nerve disease from any cause.
6. Use of systemic medications known to affect IOP (e.g., oral beta-adrenergic blockers, alpha-agonists and blockers, angiotensin converting enzyme inhibitors and calcium channel blockers), which have not been on a stable course for 7 days prior to Day 1 Visit or an anticipated change in the dosage during the course of the study.
7. A condition, which in the opinion of the Principal Investigator, would interfere with optimal participation in the study, or which would present a special risk to the subject.
8. Participation in any other investigational study within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Mean change in Intraocular Pressure (IOP) following 12 weeks of twice daily dosing | 12 weeks

SECONDARY OUTCOMES:
Percentage of subjects with IOP ≤ 18 millimeters mercury (mmHg) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mississauga, Ontario, Canada